CLINICAL TRIAL: NCT05513729
Title: Therapeutic Effects of Canagliflozin on the Liver Inflammation Damage and Lipoprotein Metabolism in Patients With Type 2 Diabetes Mellitus Combined With Nonalcoholic Fatty Liver Disease
Brief Title: Effect of Canagliflozin on Liver Inflammation Damage in Type 2 Diabetes Patients With Nonalcoholic Fatty Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2022LSK-319
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Type 2 Diabetes Mellitus With Complication
MeSH Terms: interventions — Canagliflozin; Pioglitazone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Peripheral blood samples were collected at the enrollment and the end of the study. The serum samples were separated and stored at minus 80°C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Canagliflozin treatment group: 40 patients with T2DM combined with NAFLD will be assigned to receive canagliflozin on top of metformin monotherapy according to clinical guideline of type 2 diabetes as experimental group.
  Interventions: Drug: Canagliflozin
- Pioglitazone treatment group: 40 patients with T2DM combined with NAFLD will be assigned to receive pioglitazone on top of metformin monotherapy according to clinical guideline of type 2 diabetes as experimental group. as placebo comparator group.
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Canagliflozin — According to the guideline of type 2 diabetes，canagliflozin will be given to 40 patients with type 2 diabetes combined with NAFLD as first-line choice if accompanied with indicators of high risk or established atherosclerotic cardiovascular disease, chronic kidney disease or heart failure, independently of HbA1c level. It can be also given to T2DM combined with NAFLD if their HbA1c above target.
  Other Names: Canagliflozin tablets
  Groups: Canagliflozin treatment group
Drug: Pioglitazone — According to the newest guideline of Diabetes，pioglitazone will be given to 40 patients with T2DM combined with NAFLD if their HbA1c above target.
  Other Names: Pioglitazone Hydrochloride Tablets
  Groups: Pioglitazone treatment group

SUMMARY:
Type 2 diabetes mellitus (T2DM) is always accompanied with nonalcoholic fatty liver disease (NAFLD).This prospective study was designed to reveal the potential clinical application and underlying mechanisms of canagliflozin in the treatment of type 2 diabetes combined with nonalcoholic fatty liver disease.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is one of the most important risk factors for nonalcoholic fatty liver disease (NAFLD), including nonalcoholic steatohepatitis (NASH). Thus far, there are no approved medicines to treat NAFLD/NASH and none of plasma biomarkers are sufficient to accurately and rapidly diagnose NASH in clinic. Canagliflozin is a sodium-glucose cotransporter 2 inhibitor that not only reduces glycemia, blood pressure and albuminuria, but also lowers body weight and improves dyslipidaemia. However, whether canagliflozin can be used to treat NAFLD/NASH and its impacts on lipid and lipoprotein metabolism are still rather obscure. Based on findings from our previous studies, we propose the following hypothesis: canagliflozin decreases body fat mass, in particular the visceral fat depots and liver fat content, thus alleviating hepatic steatosis, hepatic macrophage content and activation. Since we have demonstrated for the first time that plasma cholesteryl ester transfer protein (CETP) is predominantly derived from hepatic macrophages, and CETP plays a pivotal role in regulating lipid and lipoprotein metabolism. Moreover, plasma CETP concentration and activity can be applied as an effective biomarker for hepatic steatosis and liver inflammation and damage. Collectively, in this study, 80 patients with T2DM combined with NAFLD, who have been given metformin monotherapy for at least 3 months, will be assigned to receive canagliflozin or pioglitazone (as placebo control) on top of metformin according to the guideline of Type 2 diabets. The primary outcome will be plasma CETP concentration and activity, as measurements of liver lipid content, hepatic steatosis, liver inflammation and damage. The secondary outcome will be nuclear magnetic resonance spectroscopy- based metabolomics, including lipoprotein profile, lipid species and metabolomic, to comprehensively evaluate the therapeutic effects of canagliflozin on lipids and lipoproteins. We anticipate this prospective study will reveal the potential clinical application and underlying mechanisms of canagliflozin in the treatment of NAFLD/NASH, and also provide a theoretical basis for predicting its effect on cardiovascular disease events, thus having important economic value and scientific significance.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for type 2 diabetes(1999 WHO criteria).
* Meets the diagnostic criteria for non-alcoholic fatty liver disease (2018 Chinese Medical Association Treatment Guidelines ), and liver ultrasound showed moderate or higher fatty liver.
* Metformin monotherapy for 3 months
* 8 years old ≤ age ≤ 70 years old;
* Have a good follow-up compliance, with follow-up months ≥ 24 weeks;

Exclusion Criteria:

Non-type 2 diabetes: type 1 diabetes, gestational diabetes, or other specific types of diabetes;

* Diabetes patients with acute and chronic complications and serious infections; Pregnant and lactating women;
* Those who have allergies or toxic side effects or contraindications to canagliflozin, pioglitazone and other drugs;
* Active sexually transmitted diseases such as viral hepatitis, AIDS and syphilis, and infectious diseases such as tuberculosis;
* Have a weight change of more than 10% in the 3 months prior to screening;
* Have used other drugs that may affect blood glucose metabolism in the past 2 months, including systemic glucocorticoids (except inhalation or topical use), growth hormone, etc.;
* Have used any sodium-glucose cotransporter-2 (SGLT-2) inhibitor or thiazolidinediones in the 3 months prior to screening;
* History of more than 2 severe hypoglycemic episodes in the past 1 year;
* History or condition of any of the following: decompensated cardiac insufficiency (NYHA class III or IV); history of unstable angina, myocardial infarction, coronary artery bypass grafting, or coronary stenting; uncontrolled or severe heart rhythm Disorders (such as long QT syndrome, etc.), and evaluated by the investigator to be unsuitable to participate in this clinical trial; currently accompanied by clinically significant urinary tract/ reproductive infection, or a history of complicated urinary tract infection, or nearly 6 A history of recurrent urinary tract infections within a month;
* Currently known to have severe osteoporosis, or a history of secondary fractures within the past 1 year;
* Any laboratory tests meet the following criteria: fasting plasma/ serum glucose ≥ 15 mmol/L; alanine aminotransferase or aspartate aminotransferase > 3 times the upper limit of normal or total bilirubin > 1.5 times normal Upper limit; hemoglobin <100 g/L; glomerular filtration rate (eGFR) < 60 mL/min/1.73m2; fasting triglycerides > 5.64 mmol/L (500 mg/ dL);
* Has received or is receiving any other experimental drug/trial device treatment within the past 3 months;
* Other conditions deemed inappropriate by the investigator to participate in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 Diabetes Patients With Nonalcoholic Fatty Liver Disease who have been treated with metformin monotherapy for at least 3 months.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Plasma cholesteryl ester transfer protein(CETP) concentration(ug/mL) | 24 weeks after the date of enrollment
  Measurements of liver inflammation and damage
The activity of CEPT in pmol/mL/min | Time Frame: 24 weeks after the date of enrollment
  Measurements of liver inflammation and damage

SECONDARY OUTCOMES:
Plasma cholesteryl ester transfer protein(CETP) concentration in ug/mL | Baseline
  Measurements of liver inflammation and damage
The activity of CEPT in pmol/mL/min | Baseline
  Measurements of liver inflammation and damage

CONTACTS AND LOCATIONS:
Overall Officials: YAYI HE, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital Xi'an Jiaotong University, Xi'an, Shannxi, China